CLINICAL TRIAL: NCT04666103
Title: Preserving Function Integrity of Neck Anatomy in Thyroid Surgery: A Randomized Clinical Trial
Brief Title: Function Integrity of Neck Anatomy in Thyroid Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Ph D, MD, Director, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lycf202007
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Thyroid Carcinoma; Thyroid Nodule (Benign); Ablation; Retina
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroid lobectomy with intraoperative thermal ablation (Experimental): Thyroid lobectomy was performed with a standard technique of fine capsular en bloc dissection and resection, from inferior pole to superior pole. Superior parathyroid glands were identified and preserved in situ, inferior parathyroid glands were protected in situ or autotransplanted in the sternocleidomastoid muscle according to three certain types based on their blood supply and location. All the patients underwent lobectomy received ipsilateral therapic central compartment neck dissection. After the thyroid lobectomy, the contralateral benign thyroid nodule was treated with intraoperative thermal ablation. The "hydrodissection technique" was used during the ablation process to prevent recurrent laryngeal nerve, esophageal and other important structures from being destroyed by heat energy.
  Interventions: Procedure: Intraoperative thermal ablation
- Thyroid lobectomy (No Intervention): Thyroid lobectomy was performed with a standard technique of fine capsular en bloc dissection and resection, from inferior pole to superior pole. Superior parathyroid glands were identified and preserved in situ, inferior parathyroid glands were protected in situ or autotransplanted in the sternocleidomastoid muscle according to three certain types based on their blood supply and location. All the patients underwent lobectomy received ipsilateral therapic central compartment neck dissection.

INTERVENTIONS:
Procedure: Intraoperative thermal ablation — After the thyroid lobectomy, the contralateral benign thyroid nodule was treated with intraoperative thermal ablation. The "hydrodissection technique'' was used during the ablation process to prevent recurrent laryngeal nerve, esophageal and other important structures from being destroyed by heat energy.
  Arms: Thyroid lobectomy with intraoperative thermal ablation

SUMMARY:
Recent trends in the management of patients with low-risk papillary thyroid carcinoma who have a nonsuspicious or cytologically benign contralateral nodule call into question the need for routine total thyroidectomy. Although the lobectomy for the unilateral thyroid cancer with contralateral benign nodules is sufficient treatment, some of the patients might suffer from the anxiety of the residual benign thyroid nodule and tend to choose total thyroidectomy, which might be overtreatment.

Thermal ablation has been proven to be effective in achieving nodule shrinkage and being also free from major complications. In our institution, intraoperative RFA was a proposed alternative strategy to treat the contralateral benign nodules after the thyroid lobectomy for the malignant lobe, which was found to have a better quality of life on anxiety, physiological health, social family, psychological and sensory mentions with a considerable complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral thyroid carcinoma and contralateral benign nodule confirmed by preoperative ultrasound-guided fine-needle aspiration cytology;
* Patients with contralateral nodules ≤ 20mm and located in the thyroid gland;
* Patients with clinical node-negative cervical compartment at palpation and neck ultrasound.

Exclusion Criteria:

* Previous history of neck surgery
* Previous history of neck radiation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1264 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complications | Up to 2 years
  Transient or persistent hypoparathyroidism confirmed by serum calcium levels was less than the lower limit at examination center and had symptoms of hypocalcemia. Postoperative vocal cord paralysis was defined as fixed vocal cord mobility with laryngofiberoscopic examination.
Scores of hospital anxiety and depression scale (HADS) | Up to 6 months
  All patients were requested to answer the HADS questionnaire, the scores of which were recorded.
Scores of fear of progression questionnaire-short form(FPQS) | Up to 6 months
  All patients were requested to answer the FPQS questionnaire, the scores of which were recorded.
Scores of thyroid cancer- specific quality of life (THYCA-QoL) questionnaire | Up to 6 months
  All patients were requested to answer the THYCA-QoL questionnaire, the scores of which were recorded.
Rate of recurrence | 5-year estimate reported after a median follow-up of 60 months
  Lymph node recurrence or distant recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Gaosong Wu, Ph.D., Principal Investigator — Department of Breast and Thyroid Surgery, Zhongnan Hospital of Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No